CLINICAL TRIAL: NCT06819722
Title: The Effect of Parents' Health Literacy on Primary School Students' Health Screening Results
Status: Active, not recruiting | Type: Observational
Sponsor: Duzce University (Other)
Responsible Party: Sponsor
Other Study IDs: Duzce-U-merve0004
Record Dates: First submitted 2024-12-10; First posted 2025-02-11 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Health Literacy; Health Screening
Keywords: Health literacy; Health screening; Primary school students

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Parents: This group consists of parents of students studying in primary school. The Personal Information Form and the Turkey Health Literacy Scale will be completed by the parents.
- Students: This group consists of students studying in primary school. The Student General Health Form and the Student Screening Follow-up Form will be completed for the student.

SUMMARY:
Health literacy (HL) is defined by the World Health Organization (WHO) as "the achievement of a level of knowledge, personal skills, and confidence to take action to improve individual and community health by changing personal lifestyles and living conditions". Health literacy is described as a concept encompassing various skills that enhance individuals' quality of life, such as accessing accurate health information, developing healthy living behaviours, utilizing healthcare services, and making health-related decisions. To improve the health literacy of society, it is essential first to identify and enhance the health literacy of families, the smallest unit of the community. Adult family members are responsible for their health and play a critical role in fostering healthy behaviours in their children and addressing their health needs.

Aim: Health screenings, particularly for the early diagnosis of health issues in children, are crucial for health preservation and the creation of a healthy society in the future. Therefore, the aim of this study is to determine the health literacy of parents and its impact on the health screening results of students.

DETAILED DESCRIPTION:
Health literacy (HL) is defined by the World Health Organization (WHO) as "the achievement of a level of knowledge, personal skills, and confidence to take action to improve individual and community health by changing personal lifestyles and living conditions". Health literacy is a concept encompassing various skills that enhance individuals' quality of life, such as accessing accurate health information, developing healthy living behaviours, utilizing healthcare services, and making health-related decisions. To improve the health literacy of society, it is essential first to identify and enhance the health literacy of families, the smallest unit of the community. Adult family members are responsible for their health and play a critical role in fostering healthy behaviours in their children and addressing their health needs. It is also known that parents act as role models in developing children's positive health behaviours and enhancing their quality of life. Low health literacy is known to be associated with negative health outcomes in adults. In this context, it is stated that parents who struggle to take responsibility for their health may also face difficulties in meeting their children's health needs, and consequently, inevitably, children frequently encounter health problems. Studies have found that parents with low health literacy struggle with meeting their children's health needs, using healthcare services, taking preventive measures against health risks, proper medication use and monitoring side effects, managing chronic diseases, and encouraging their children to adopt healthy living behaviours. In particular, during the school-age period, which is one of the critical periods for the healthy and successful development of society, as children rapidly develop socially, physically, and cognitively, it is stated that early detection of children's health needs and problems by their parents and the timely receipt of necessary health services can prevent more serious problems that may arise later. In Turkey, recently, the continuous monitoring of the health of schoolchildren, early detection of health risks, and the continuity of practices aimed at promoting health was addressed by the Ministry of National Education, which published the "Regulations on the Working Procedures and Principles of School Health Nurses" on 20/04/2020. As a result, school health nurses have been employed by this regulation. Under the "Regulation on the Amendment of the Nursing Regulation" published by the Ministry of Health in 2011, school health nursing, which is a dimension of public health nursing, includes health screenings as one of the practices that can be carried out independently. Health screenings are crucial for the early diagnosis of children's health problems, health preservation, and the creation of a healthy society in the future. Therefore, the aim of this study is to determine the health literacy of parents and its impact on the health screening results of students. It is believed that the study could contribute to the development of health services and policies aimed at increasing public health and health literacy, preventing health inequalities, and increasing the visibility of school health nursing activities, which are becoming increasingly important. This, in turn, would contribute to the protection and improvement of both parental and child health.

ELIGIBILITY:
Inclusion Criteria:

* Students and parents attending Sancaklar Primary School located in Düzce city centre.
* Voluntary participation in the study.

Exclusion Criteria:

* Parents who do not agree to participate in the study and their children will be excluded from the research.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The research will be conducted at Sancaklar Primary School, located in the centre of Düzce, between September 2024 and June 2025. A total of 188 students and their parents attending Sancaklar Primary School will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 376 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Health literacy | one day
  The Turkey Health Literacy Scale was developed by Okyay and Abacıgil in 2016 to assess health literacy, in line with the European Health Literacy Research Consortium. The scale consists of 32 questions. It has a 2x4 matrix structure, with two dimensions (treatment and services, and disease prevention/health promotion) and four processes (accessing health-related information, understanding health-related information, evaluating health-related information, and using/applying health-related information), making a total of eight components. The Cronbach's Alpha value of the scale is 0.927. The scale is rated as follows: "1. Very Easy, 2. Easy, 3. Neither easy nor difficult, 4. Difficult, 5. Very Difficult." The health literacy level is categorized into four groups based on the score obtained: (0-25) points: Inadequate health literacy, (>25-33) points: Problematic - limited health literacy, (>33-42) points: Adequate health literacy, (>42-50) points: Excellent health literacy.
Health Screening (Height) | From March 2025 to May 2025
  The height (m) of primary school students will be measured by meter
Health Screening (Weight) | From March 2025 to May 2025
  Primary school students' weight (kg) will be measured by scales
Health Screening (Body Mass Index) | From March 2025 to May 2025
  Body mass index (kg/m^2) will be calculated after weight and height measurement.
Health Screening (The temperature) | From March 2025 to May 2025
  The temperature of primary school students will be measured with a thermometer
Health Screening (Pulse rate) | From March 2025 to May 2025
  The pulse rate per minute (beats/min) of primary school students will be measured.
Health Screening (The respiratory rate) | From March 2025 to May 2025
  The respiratory rate per minute of primary school students will be measured.
Health Screening (Blood Pressure) | From March 2025 to May 2025
  Primary school students' blood pressure will be measured with child-friendly blood pressure monitors.
Health Screening (Oral and Dental Health Screening) | From March 2025 to May 2025
  Oral and dental health screenings will be conducted for primary school students.
Health Screening (Hair, Ear and Nail Evaluation) | From March 2025 to May 2025
  Hair, ear and nail health screenings will be conducted for primary school students.
Health Screening (Scabies) | From March 2025 to May 2025
  Primary school students will be screened for scabies.
Health Screening (Eye Screening) | From March 2025 to May 2025
  Eye screening of primary school students will be done using Snellen and Snellen E charts.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Cakar, PhD, Principal Investigator — Duzce University
Locations (1):
- Duzce University, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No